CLINICAL TRIAL: NCT00200577
Title: TIL (Tumor Infiltrating Lymphocytes) and IL2 (Interleukin 2) Versus Abstention as Adjuvant Treatment in Melanoma With Only One Invaded Lymphnode After Lymphnodes Excision
Brief Title: Tumor Infiltrating Lymphocytes Adjuvant Therapy of Melanoma
Acronym: TIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/04/01-D
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Melanoma
Keywords: Adjuvant therapy; immunotherapy; TIL; melanoma
MeSH Terms: conditions — Melanoma | interventions — Toll-Like Receptor 1; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIL+IL2 (Experimental): TIL + IL2
  Interventions: Drug: TIL + IL2
- control (No Intervention): Patients are not treated

INTERVENTIONS:
Drug: TIL + IL2 — Patients are treated with 2 injections Of TIL (1st injection M1 and the second M2)The received concomitant IL2 at M1 and M2 on days Jo (injection TIL) to J5 and J8 to J12
  Arms: TIL+IL2

SUMMARY:
The objective of this multicentric Phase III study is to confirm the results of the phase I-II study (Dreno B & Al. Cancer Immunol Immunother 2002; 51: 539-456) which demonstrated the preventive effect of a treatment by TIL (Tumor Infiltrating Lymphocytes) combined with IL2 (Interleukin 2; low dose injected subcutaneously) on the metastatic relapse in the stage III melanoma patients with only one invaded lymphnode.

DETAILED DESCRIPTION:
In this open, multicentric (Grenoble, Montpellier, Nantes, Angers, Caen, Le Mans, Poitiers, Rennes, Tours) randomized study, selected patients with only one invaded lymphnode confirmed by anatomopathological exam will be randomized to one of the following arms: 1-Control group: patients of this group will not receive any treatment and will have the same clinical follow-up as the treated group. 2- TIL-IL2 group: treated patients will receive two injections of TIL combined with IL2. Tumor Infiltrating Lymphocytes will be obtained from a small piece of tumour tissue removed from the invaded lymphnode after surgery. TIL will be grown in larger number in laboratory during 6 weeks. Patients randomized in treatment arm will receive two injection of TIL (the first about 6 and the second about 10 weeks post-surgery). Administration of TIL will be combined with a low dose of IL2 (6 million U.I. per day) injected subcutaneously from J1 to J5 and J8 to J12 following the day of TIL infusion. The same dose and duration of IL2 treatment will be used for the second injection of TIL performed one month later. After 2 months adjuvant therapy, patients received no other treatment. Only a regular follow-up was performed.

ELIGIBILITY:
Inclusion Criteria:

* Melanoma stage III (regional lymph node recurrence). Will be selected the patients with only one invaded lymph node confirmed by anatomopathological exam after lymph nodes excision.
* Absence of visceral metastases verified by physical examination, chest radiography, liver echography and brain-chest-liver CT-Scan.
* Age < 75 years, both genders
* ECOG 0-2, Karnofsky > 80%.
* Negative pregnancy test performed at the screening visit for fertile women.
* The potentially fertile women must use an oral contraception or an intra-uterine device (IUD) until three months following the last injection of the study treatment.
* The patients must have fully recovered from surgery.
* HIV 1/2: The patients must be negative for antibodies HIV 1 and HIV 2 and for Ag P24 or DGV HIV.
* HBV: The patients must be negative for the antigen, but can be positive for the antibodies but with a negative DNA PCR.
* HCV: The patients must be negative for the antibodies.
* HTLV ½: The patients must be negative for the antibodies.
* Following laboratory results:

  * Hemoglobin: ≥ 10 g/dl
  * WBC: ≥ 4000/µl
  * Lymphocytes: ≥ 700/µl
  * Platelet count: ≥ 100.000/µl
  * Serum creatinine: < 2.0 mg/dl or £ 177 mmol/l
  * Serum Bilirubin: < 2.0 mg/dl or £ 34.2 mmol/l
  * ASAT and ALAT: < 2.5 x the upper limit of normal.

Exclusion criteria:

* Patient with more than one invaded lymph node confirmed by anatomopathological exam.
* Presence of melanoma metastases discovered by clinical or radiological examination at the screening visit.
* Patients must not have received any Chemotherapy, immunotherapy or radiotherapy within the preceding 4 weeks (6 weeks since prior nitrosurea and mitomycin C therapies).
* Presence of cardiac affections (congestive cardiac insufficiency, coronaropathy, not controlled HTA).
* Any serious active medical illnesses, for example: Active systemic infections requiring of antibiotics, coagulation disorders or any other condition which requires concomitant medications not allowed during this study.
* Presence of the second active cancer other than surgically cured non-melanoma skin cancer or cervical carcinoma in-situ.
* Any affection requiring a systemic corticotherapy or a treatment by Interferon A.
* Any active auto-immune disease including the insulin-dependent diabetes or a immunodeficiency. The vitiligo is not an exclusion criteria.
* Thyroid dysfunction not responsive to therapy.
* Positive Serology for HIV, HVB, HVC or HTLV1/2.
* Woman pregnant or nursing or without an effective contraception.
* Incapacity to give written consent.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Determination of the duration of the relapse-free interval. | 5 years
Physical examination, every 2 months until M18 then every 3 months until M36 then every 4 months up to 5 years, then once per year with a clinical examination only. | every 2 months until M18then every 3 months until M36 then every 4 months up to 5 years
Abdominal echography will be performed at the screening visit, M4, M8, M12 and then every 6 months until 5ans. | M4, M8, M12 and then every 6 months until 5ans.
CT-Scan will be performed before the first administration of study treatment (at the time of screening visit), every 6 months during 2 years and then every years up to 5 years. | every 6 months during 2 years and then every years up to 5 years.

SECONDARY OUTCOMES:
Determine of overall survival | 5 years
To define safety and toxicity of TIL/IL2 treatment | 5 years
Evaluation of immunological responses | M0, J56, M12
Analysis of the clinical, biological and histological factors on the survival of the patients | at inclusion and each month

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte DRENO, MD, Principal Investigator — Nantes University Hospital
Locations (9):
- France (9):
  - CHU Angers, Angers
  - CHU Caen, Caen
  - Grenoble University Hospital, Grenoble
  - CH Le Mans, Le Mans
  - Montpellier University Hospital, Montpellier
  - Nantes University Hospital, Nantes
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHRU Tours, Tours